CLINICAL TRIAL: NCT05709158
Title: Evaluation of Risk Factors Associated With Myelosuppression (Grade 4 Neutropenia) in Breast Cancer Patients Treated With Palbociclib in the Post-marketing Setting: Nested Case-control Study Using the Medical Information Database Network (MID-NET) Database
Brief Title: A Study to Learn About the Dangers Linked to Myelosuppression (Decreased Bone Marrow Function) in Breast Cancer Patients Treated With the Study Medicine Palbociclib (Pal Bow Sai Klib)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481093
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
Keywords: Safety; data base study in Japan; Ibrance; Palbociclib; hormone receptor-positive (HR+)/human epidermal growth factor receptor 2-negative (HER2-); inoperable or recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

GROUPS / COHORTS (2):
- Case: G4 neutropenia occurs after palbociclib initiation: Grade 4 neutropenia occurs after initiation of palbociclib Note that: Case patients are categorized as control before incurring grade 4 neutropenia
- Control: G4 neutropenia does not occur after palbociclib initiation: Grade 4 neutropenia does not occur after initiation of palbociclib

SUMMARY:
The purpose of this study is to explore risk factors for grade 4 neutropenia in users of the study medicine Palbociclib for the potential treatment of Palbociclib.

This study is seeking participants:

* treated with the study medicine Palbociclib
* having any breast cancer records in same month as the initiation date
* having prescription records of palbociclib from 15 December 2017 to 29 February 2024

The study design is a nested case control study. This study design uses de-identified patient data from a hospital based electronic medical record and claim database in Japan. This design was selected since the primary objective is to explore risk factors of Grade 4 neutropenia in users of the study medicine Palbociclib.

One of the important side effects of taking Palbociclib is neutropenia (decreased count of neutrophils - a type of white blood cell).

In this study the effect of Palbociclib in decreasing the neutrophil count was studied after it was released to the market.

To do that, the study gathered details of breast cancer patients newly treated with Palbociclib from 23 hospitals and 10 medical institutes across Japan.

The below patient details were collected:

* dose of Palbociclib
* other medicines prescribed for cancer
* age
* gender
* past information on cancer treatments
* laboratory findings at baseline

The result was based on the neutrophil count collected from the laboratory data.

Around 1300 patients newly treated with Palbociclib for breast cancer was calculated by the medical information database network (MID-NET) in 6 years from 15 December 2017.

Patients who develop grade 4 neutropenia after palbociclib initiation will be matched to controls who do not develop grade 4 neutropenia. A statistical model will be used to explore risk factors of grade 4 neutropenia adjusted for important potential confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* Having prescription records of palbociclib from 15 December 2017 to 29 February 2024.
* Having any breast cancer records in same month as the first prescription date.

Exclusion Criteria:

* Having an ANC less than the threshold value for grade 4 neutropenia within 30 days of the first prescription of palbociclib
* Having any records of anti-HER2 medication

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Breast cancer patients treated with Palbociclib
Sampling Method: Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Risk Factors for Grade 4 Neutropenia in Users of Palbociclib | 01 Jun 2017 through 29 Feb 2024
  Grade 4 neutropenia, as the outcome of this study, will be defined as an absolute neutrophil count (ANC) of less than 0.5 × 109 cells/L or less than 500 cells/mL during the "on-treatment" period.

SECONDARY OUTCOMES:
Number of Participants With Risk Factors for Grade 4 Neutropenia in New Users of Palbociclib | 20 Dec 2016 through 29 Feb 2024
  Grade 4 neutropenia, as the outcome of this study, will be defined as an ANC of less than 0.5 × 109 cells/L or less than 500 cells/mL during the "on-treatment" period.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481093